CLINICAL TRIAL: NCT04310865
Title: An Adaptive, Randomized, Double-blind, Parallel-controlled Clinical Trial of Yinhu Qingwen Granula for the Treatment of Severe CoVID-19
Brief Title: Yinhu Qingwen Granula for the Treatment of Severe CoVID-19
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: There were no eligible patients with CoVID-19 in the paticipated centers.
Sponsor: Zhong Wang (Other)
Collaborators: Wuhan Leishenshan Hospital (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); Tanshan People's Hospital (Unknown); North China University of Science and Technology (Other); Jizhong Energy Fengfeng Group Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YHQW-Severe-V2.0
Record Dates: First submitted 2020-03-15; First posted 2020-03-17 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Severe Pneumonia; Chinese Medicine
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yinhu Qingwen Granula Group (Experimental): Based on the standard medical treatment, the patients will be given Yinhu Qingwen Granula for 10 days.
  Interventions: Drug: Yinhu Qingwen Granula; Other: standard medical treatment
- Yinhu Qingwen Granula Low-dose Group (Placebo Comparator): Based on the standard medical treatment, the patients will be given 10% dose of Yinhu Qingwen Granula for 10 days.
  Interventions: Drug: Yin Hu Qing Wen Granula(low does); Other: standard medical treatment

INTERVENTIONS:
Drug: Yinhu Qingwen Granula — Yinhu Qingwen Granula is a kind of herbal granula made from "Yinhu Qingwen Decoction", which consits of 11 Chinese herbal medicine as Honeysuckle, Polygonum cuspidatum, Schizonepeta, Longspur epimedium, etc. The granula will be dissolved into 600ml decoction and divided to 3 times (once with 200ml). It will be given a 200ml per time, three times a day, for 10 days.
  Arms: Yinhu Qingwen Granula Group
Drug: Yin Hu Qing Wen Granula(low does) — This intervention is given as 10% dose of YinHu QingWen Granula.The granula will be dissolved into 600ml decoction and divided to 3 times (once with 200ml).
  Arms: Yinhu Qingwen Granula Low-dose Group
Other: standard medical treatment — Standard medical treatment is adhered to the protocol of the treatment for the severe CoVID-19 according to the guideline approved by National Health Commission of China.

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia caused by CoVID-19, and the number of cases of infection with CoVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally.Given no specific antiviral therapy for CoVID-19 infection and the availability of Yinhu Qingwen Granula as a potential antiviral Chinese medicine based on vivo antiviral studies in CoVID-19, this adaptive, randomized,double-blind,controlled trial will evaluate the efficacy and safety of Yinhu Qingwen Granula in patients hospitalized with severe CoVID-19.

DETAILED DESCRIPTION:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia caused by CoVID-19, and the number of cases of infection with CoVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally.The clinical spectrum of CoVID-19 infection appears to be wide,including asymptomatic infection, mild upper respiratory disease, severe viral pneumonia with respiratory failure, and even death. However,there is no specific antiviral therapy for CoVID-19 infection, which provides a window of opportunity for testing candidate antiviral therapies. Previous experiences with SARS and MERS-CoV, highlight the need of the early intervention with Chinese medicine, and so as for CoVID-19 infection. The treatment of Chinese medicine for CoVID-19 infection suggested its benefits to improve of clinical outcomes, reduce the risk of disease progression, accelerate recovery, and reduce intensive supportive care and long-term hospitalization.Yinhu Qingwen Granula was a kind of herbal granula made from "Yinhu Qingwen Decoction", which consists of 11 common non-toxic traditional Chinese medicine such as Polygonum cuspidatum, Honeysuckle, Nepeta, Ligustrum lucidum. Previous vivo antiviral studies showed its activity for the inbition of CoVID-19. This clinical trial is planned to evaluate the improvement of the changes in the ratio of PaO2 to FiO2 from the baseline for patients with severe CoVID-19 as the primary outcome, and to evaluate the effect of the symptoms relief and virus clearance as well as the clinical safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of signing Informed Consent Form;
2. Those who meet the diagnosis of severe new coronavirus pneumonia with laboratory confirmed infection with CoVID-19;
3. Lung involvement confirmed with chest imaging;
4. Hospitalized with a Pa02/Fi02 ratio ≤300mgHg;
5. 40%> lymphocyte percentage ≥5%;
6. No difficulty swallowing oral medications.

Exclusion Criteria:

1. Allergies, those who are known to be allergic to research drugs or drug excipients;
2. The patient weighs less than 40 kg;
3. Patients with diarrhea;
4. Shock;
5. Patients with respiratory failure at the time of enrollment who need invasive mechanical ventilation;
6. The clinician judges that ICU admission is needed;
7. Patients who participated in other clinical trials within 1 month;
8. Known patients with impaired renal function (estimated creatinine clearance <60 mL / min (male: Cr (ml / min) = (140-age) × body weight (kg) / 72 × blood creatinine concentration (mg / dl); female: Cr (ml / min) = (140-age) × weight (kg) / 85 × blood creatinine concentration (mg / dl));
9. During the screening or within 24 hours before screening, patients were found to have any of the following laboratory parameter abnormalities (based on the local laboratory reference range): ALT or AST level> 5 times the upper limit of normal range (ULN) or ALT or AST level> 3 times ULN and total bilirubin levels> 2 times ULN;
10. Being pregnant or breastfeeding, or having a positive pregnancy test at the time of pre-dose inspection, or planning to become pregnant within 3 months after study treatment;
11. Will be transferred to another hospital which is not the study site within 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
changes in the ratio of PaO2 to FiO2 from baseline | Day 10

SECONDARY OUTCOMES:
PaO2 | up to 30 days
blood oxygen saturation (SpO2) | up to 30 days
clinical status rating on the 7-point ordinal scale | up to 30 days
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Time to Clinical Improvement (TTCI) | up to 30 days
  TTCI is defined as the time (in days) from initiation of study treatment (Yinhu Qingwen Granula or its low-dose granula) until a decline of two categories from status at randomisation on the 7-point ordinal scale of clinical status which ranges from 0 (death) to 6 (Not hospitalized, no limitations on activities).
Duration (hours) of non-invasive mechanical ventilation or high-flow nasal catheter oxygen inhalation use | up to 30 days
Duration (hours) of invasive mechanical ventilation use | up to 30 days
Duration (hours) of extracorporeal membrane oxygenation (ECMO) use | up to 30 days
Duration (days) of Oxygen use | up to 30 days
The proportion of the patients reporting 2019-nCoV RT-PCR negativity at Day 10 after treatment | Day 10
The counts/percentage of Lymphocyte | up to 30 days
Time to hospital discharge with clinical recovery from the randomisation | up to 30 days
The incidence of critical status conversion in 30 days | up to 30 days
  Critical status is defined as: 1) respiratory failure with the need of invasive mechanical ventilation; or 2) shock; or 3) other system organ failure with ICU admission.
All-cause mortality within 30 days | up to 30 days
Frequency of severe adverse drug events | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dong Shang, M.D., Principal Investigator — Wuhan Leishenshan (Thunder God Mountain) Hospital/The First Affiliated Hospital of Dalian Medical University; Jiang-Rong Huang, M.D., Principal Investigator — Yangtze University Health Science Center; Xiao-Dong Li, M.D., Principal Investigator — Hubei Hospital of Traditional Chinese Medicine; Zhong Wang, M.D., Study Director — China Academy of Chinese Medical Sciences
Locations (4):
- China (4):
  - Wuhan No.7 Hospital/Jizhong Energy Fengfeng Group Hospital, Wuhan, Hubei
  - Wuhan No.7 Hospital/North China University of Science and Technology Affiliated Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University/Tanshan People's Hospital, Wuhan, Hubei
  - Wuhan Leishenshan (Thunder God Mountain) Hospital/The First Affiliated Hospital of Dalian Medical University, Wuhan, Hubei